CLINICAL TRIAL: NCT02813187
Title: A Real World, Observational Registry of Venous Leg Ulcers and Quality of Care in Clinical Practice
Brief Title: Venous Leg Ulcer and Lymphedema Registry
Acronym: VLULR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: U.S. Wound Registry (Other)
Responsible Party: Sponsor
Other Study IDs: CDR006
Record Dates: First submitted 2016-06-10; First posted 2016-06-24 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Venous Stasis Ulcer; Quality of Patient Care
Keywords: venous leg ulcer; venous; QCDR; quality measure; wound; Outcome; Lymphedema
MeSH Terms: conditions — Varicose Ulcer; Wounds and Injuries; Lymphedema | interventions — Cell Count; Apligraf; TransCyte; Debridement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cellular and tissue based therapy
  Other Names: Apligraf; Dermagraft; Theraskin; Epifix; Dermapure; Grafix; Talymed
Procedure: debridement
Procedure: advanced wound therapy
Dietary Supplement: Nutritional screening

SUMMARY:
This is an observational, longitudinal real world registry of venous leg ulcers created from electronic health record data obtained in the course of clinical care. Data from certified electronic health records transmit data as part of the requirement to share data with a specialty registry under Objective 10 of Meaningful Use of an EHR.

DETAILED DESCRIPTION:
This is an observational, longitudinal real world registry of venous leg ulcers created from electronic health record data obtained in the course of clinical care. Data from certified electronic health records transmit data as part of the requirement to share data with a specialty registry under Objective 10 of Meaningful Use of an EHR. No secondary data entry are required and all data are obtained via structured language from data entered in the EHR. Data from quality measures designed as electronic clinical quality measures (eCQMs) standardize the quality of care provided to patients and their clinical outcomes which are risk stratified using the Wound Healing Index (WHI). The eCQMs enable standardized data collection and the ability to transmit data electronically obviates the possibility of transcription errors. National bench marking is possible since data are available from thousands of participants across the USA. While an independent IRB oversees this project, the data are collected for the purpose of measuring and improving the quality of care delivered to diabetic patients with foot ulcers and understanding their outcomes in relation to level of risk. Quality performance is reported as part of PQRS. These functions are exempt from the requirements of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* All patients with venous leg ulcers seen by the practitioner.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospectively followed venous leg ulcers in the practice of clinicians submitting data to the registry
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 12 months
  wound closure

SECONDARY OUTCOMES:
Weeks of Therapy | 12 months
  days from initial visit to discharge
Adverse events during therapy | 12 months
  hospitalization, cellulitis, amputation
Patient Reported Outcome | 12 months
  using patient reported outcome quality measure
Venous Insufficiency | 12 months
  secondary lymphedema and its relationship to venous insufficiency

CONTACTS AND LOCATIONS:
Locations (1):
- CHI St. Luke's The Woodlands, The Woodlands, Texas, United States